CLINICAL TRIAL: NCT02327663
Title: Emtricitabine for Naive Chinese Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asian-Pacific Alliance of Liver Disease, Beijing (Other)
Collaborators: Beijing Ditan Hospital (Other); Hebei Medical University Pharmaceutical Factory (Industry); National Health and Family Planning Commission, P.R.China (Other Government)
Responsible Party: Principal Investigator, Jun Cheng, chaireman of Asian-Pacific Alliance of Liver Diseas,Beijing, Asian-Pacific Alliance of Liver Disease, Beijing
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FTC-01
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, chronic; Emtricitabine; Adefovir dipivixil; HBeAg
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HBeAg positive CHB group (Experimental): 1000 patients take generic emtricitabine capsule(200 mg one time per day) for 96 weeks,and for patients who have HBV DNA > 500 copies/ml, adefovir dipivoxil were combined
  Interventions: Drug: Emtricitabine
- HBeAg negativie CHB group (Experimental): 1000 patients take generic emtricitabine capsule(200 mg one time per day) for 96 weeks,and for patients who have HBV DNA > 500 copies/ml, adefovir dipivoxil were combined
  Interventions: Drug: Emtricitabine

INTERVENTIONS:
Drug: Emtricitabine — emtricitabine were given to each patients at baseline and respoonse guided therapy was adopted according HBV DNA level at week 24
  Other Names: Brand name：Huierding

SUMMARY:
This study evaluates generic emtricitabine(FTC) in Chinese naive chronic hepatitis B patients. Patients were divided into 2 groups: HBeAg positive Chronic hepatitis B(CHB)group and HBeAg negative Chronic hepatitis B(CHB)group.

DETAILED DESCRIPTION:
Generic emtricitabine(FTC) has been approved for treatment of naive chronic hepatitis B(CHB) patients in China. Yet data are limited for this agent. The investigators design this trial to test the effect of FTC in Chinese CHB which including naive HBeAg positive and Negative CHB patients. Response guided therapy strategy is adopted for patients who can not achieve HBV DNA negativity at week 24 FTC treatment, which means FTC and adefovir are combined for these patients.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive for more than 6 months
* HBeAg positive patients: HBV DNA ≥ 5log10 copies/ml
* HBeAg postive patients: ALT≥2×ULN;or liver biopsy G≥2;or liver biopsy S ≥2;or liver biopsy Knodell HAI ≥ 4
* HBeAg negative patients: HBV DNA ≥ 4log10 copies/ml
* HBeAg postive patients: ALT≥2×ULN;or liver biopsy G≥2;or liver biopsy S ≥2;or liver biopsy Knodell HAI ≥ 4
* nucleoside/nucleotide naive paitents

Exclusion Criteria:

* Diagnosed HCC with AFP and ultrasound, CT or MRI
* Creatine >130μmol/L or Ccr < 70mL/min
* Hemoglobin <100g/L
* Neutrophils <1.5E+9/L
* PLT<80E+9/L
* Coinfected with HAV,HEV,HCV,HDV or HIV
* ANA > 1:100
* Uncontrolled cardiovascluar diseases, kidney diseases,lung diseases, neurological diseases, digestive diseases,metabolic disorders, immune-compromised diseases or cancer
* Drug abuse or alcohal addiction
* Previous history of taking agents of lamivudine, adefovir, tenofovir entecavir or telbivudine
* Long-term use of immunosuppressor or immunomodulator 6 months before enrollment to this trial
* Underwent liver transplantation or liver transplantation in schedule
* Allergic to nucleoside or nucleotide analogues
* Preganency or in breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
virological response rate | week 96
  HBV DNA < 500 copies/ml

SECONDARY OUTCOMES:
HBV DNA decrease level | week24, 48, 72 and 96
  HBV DNA decrease compared with baseline（log10 copies/ml）
HBV DNA negativity rate | week 24, 48 and 72
  HBV DNA < 500 copies/ml
biochemical response | week 24,48,72 and 96
  ALT normalization
HBeAg loss | week 24,48,72 and 96
  HBeAg loss in HBeAg positive group
HBeAg seroconversion | week 24,48,72 and 96
  HBeAg seroconversion in HBeAg positive group
HBeAg reversion | week 24,48,72 and 96
  HBeAg positive in Baseline HBeAg negativie group patients
HBsAg loss | week 24,48,72 and 96
  HBsAg loss in both group
HBsAg seroconversion | week 24,48,72 and 96
  HBsAg loss and anti-HBs positive
adverse event | week 24,48,72 and 96
  type and rate of adverse events;type and rate of severe adverse event;
HBV genetic resistance to emtricitabine and adefovir | week 24,48,72 and 96
  HBV genetic resistance to emtricitabine and adefovir

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cheng, M.D., Principal Investigator — Asian Pacific Alliance of Liver Diseases, Beijing

REFERENCES:
- [Background] Lim SG, Ng TM, Kung N, Krastev Z, Volfova M, Husa P, Lee SS, Chan S, Shiffman ML, Washington MK, Rigney A, Anderson J, Mondou E, Snow A, Sorbel J, Guan R, Rousseau F; Emtricitabine FTCB-301 Study Group. A double-blind placebo-controlled study of emtricitabine in chronic hepatitis B. Arch Intern Med. 2006 Jan 9;166(1):49-56. doi: 10.1001/archinte.166.1.49. PMID 16401810
- [Result] Gish RG, Leung NW, Wright TL, Trinh H, Lang W, Kessler HA, Fang L, Wang LH, Delehanty J, Rigney A, Mondou E, Snow A, Rousseau F. Dose range study of pharmacokinetics, safety, and preliminary antiviral activity of emtricitabine in adults with hepatitis B virus infection. Antimicrob Agents Chemother. 2002 Jun;46(6):1734-40. doi: 10.1128/AAC.46.6.1734-1740.2002. PMID 12019083